CLINICAL TRIAL: NCT04377763
Title: Developement and Evaluation of Serological Assays for COVID-19
Acronym: SEROCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 20MWI-SEROCOV
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: COVID-19; serological assay
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study aims to evaluate serological assays of virus Covid-19.

DETAILED DESCRIPTION:
This is a retrospective monocentric study, which will include the patients who have hospitalized in Ambroise Paré Hospital and have sampling sent to the Laboratory of Microbiology of the hospital between the 15 March 2020 and 30 september 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years;
* Have molecular diagnosis of positive or negative result in Covid-19 virus by the Laboratory of Microbiology in Ambroise Paré Hospital;
* Have diagnosed of a viral infection in respiratory.

Exclusion Criteria:

- Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with positive or negative molecular diagnosis of Covid-19, in the Laboratory of Microbiology of Ambroise Paré Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Sensibility and specificity | Throughout of the study, an average of 6 months
  Determination of sensibility and specificity of serological testing in SARS-CoV-2 virus in patients with acute respiratory symptoms.

SECONDARY OUTCOMES:
Delay between the first symptoms and the positive serological result | Throughout of the study, an average of 6 months
  Delay between the first symptoms and the positive serological result of SARS-CoV-2 virus.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Anne RAMEIX-WELTI, MD, PhD, Principal Investigator — Laboratoire de Microbiologie Hygiène hospitalière, Hôpital Ambroise paré, APHP
Locations (1):
- Laboratory of microbiology of hospital hygiene, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No